CLINICAL TRIAL: NCT03689621
Title: Proof of Concept Study of Vagus Nerve Stimulation Using an External Device for the Treatment of Behaviour Problems in People With Neurodevelopmental Disorders, Specifically Prader Willi Syndrome
Brief Title: Proof of Concept Study of Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Beresford-Webb (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Sponsor-Investigator, Jessica Beresford-Webb, Research Assistant, University of Cambridge
Organization: University of Cambridge (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15/EE/0450
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Transcutaneous Vagal Nerve Stimulation (tVNS); Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous vagal nerve stimulation (tVNS) (Active Comparator): tVNS administered for 4 hours each day and behaviour is recorded.
  Interventions: Device: Transcutaneous vagus nerve stimulation (tVNS)
- Baseline (Placebo Comparator): tVNS worn but not switched on whilst collecting behavioural data.
  Interventions: Device: Transcutaneous vagus nerve stimulation (tVNS)

INTERVENTIONS:
Device: Transcutaneous vagus nerve stimulation (tVNS)

SUMMARY:
The investigator's recent pilot study of vagus nerve stimulation (VNS) from a surgically implanted medical device to control the excess eating behaviour characteristic of Prader-Willi Syndrome (PWS) found that it was safe and acceptable. In addition, there were unanticipated marked improvements in rates of problem behaviours, such as emotional disturbances and verbal and physical outbursts. These observations indicated the need for a trial specifically focusing on the effects of VNS on problem behaviour and also that the use of VNS might be extended to include people with other neurodevelopmental disorders, such as autism spectrum conditions (ASC). The primary aims of this study are: a) to investigate whether VNS, now given by an external medical device, is associated with a significant reduction in the number and severity of maladaptive behaviours in adults with PWS; and b) to undertake a pilot study that includes others with a different neurodevelopmental syndrome who have histories of similar behaviours.

The study will be a single case cross-over design with 4 to 6 months baseline phase and a similar period of active treatment. The study cannot be blind as the stimulation is apparent but the participants will wear the device initially for four hours a day, at times convenient to them, with it switched off in the baseline phase and activated, according to standard protocols, in the treatment phase. Six adults with PWS and six with a different neurodevelopmental disorder with histories of significant problem behaviours will be included initially, with a view to extending if the analysis indicates a likely effect. Behaviours will be operationally defined and measured over time using participant and informant diaries with additional secondary outcome measures. Before and during the treatment phases autonomic nervous system and brain biomarkers will be assessed using ambulatory monitoring of heart rate variability and fMRI brain scans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged over 18 years of age.
* Genetically and clinically determined diagnosis of PWS or meeting clinical or the presence of another neurodevelopmental syndrome such as an autistic spectrum condition.
* History of problem behaviours of, on average, at least one significant informant-reported episode each week.
* Capacity to consent.
* Able to commit to the study duration and to attend assessments in Cambridge.

Exclusion Criteria:

* Meet exclusion criteria for MRI scanning and/or unable to tolerate MRI environment.
* Serious co-morbid physical or psychiatric disorder which would disrupt ability to comply with study demands (e.g. a history of serious bipolar disorder; sleep apnoea not well-controlled with CPAP; insulin dependent diabetes).
* Current or past history of neurological disorders or trauma, including epilepsy, and head injury.
* Currently or recently (within 12 months) participating in a clinical trial of an investigational medicinal product (CTIMP) or another medical device.
* Lacking the capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The number of operationally defined outbursts | 15-17 months
  Measured using participant and informant diaries.

SECONDARY OUTCOMES:
The Challenging Behaviour Checklist | 15-17 months
  Scores on rating scale, repeated over time. Score range 50-55. higher score indicates more severe behaviour.
Repetitive Behaviour Questionnaire | 15-17 months
  Scores on rating scale, repeated over time. Total scores range between 20-60. The higher toe score the worse behaviours are.
Life Experiences Checklist. | 15-17 months
  Intended to gather information about the potentially traumatic experiences a person has experienced. There is no formal scoring protocol or interpretation per se, other than identifying whether a person has experienced one or more of the events listed. Respondents indicate varying levels of exposure to each type of potentially traumatic event included on a 6-point nominal scale, and respondents may endorse multiple levels of exposure to the same trauma type.
fMRI at resting and on-task | 15-17 months
  FMRI data will be analysed using both 1st and 2nd level general linear model (GLM) analyses to compare within cases and across time points. Network analyses of functional connectivity may also be appropriate
Participants response to challenge | 15-17 months
  Using methodology developed by Prof Oliver, filmed and subsequently rated blind for emotional and behavioural changes.
Semi-structured interviews | 15-17 months
  With participants and carers to probe about any observed subtle changes in behaviour. Analysed thematically.
Attention shifting ability | 15-17 months
  Tested via go-no-go task developed for people with PWS by Woodcock et al (2009). Reaction times analysed.
Salival cortisol measures | 15-17 months
  recorded across the course of four separate days during the course of study (at waking, 30 minutes post-waking, 45 minutes post-waking, 1 hour post-waking and then four more times throughout the day at approximately +3h, +6h, +9h and +14h after waking).
Vocal prosody | 15-17 months
  Two voice recordings of the participant talking will be collected on each of these occasions. Each recording will be at least 20 seconds long, with the participant asked to talk about a positive experience (e.g. favourite birthday, best friend etc.) in one, a less positive time (e.g. a time when he/she was disappointed or sad) in the other. These will be analysed for changes in vocal prosody with t-VNS.
Heart Rate Variability | 15-17 months
  derived from ECG and respiration measured using an Intelesens (Belfast) 3-axis 'Zensor' wearable monitor. For each participant ECG recording will take place in 24-hour blocks. HRV will be determined from R-R intervals as root mean of squared successive differences and average HRV will be determined for each participant for brief (15 minutes) and prolonged (24 hours) periods.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Holland, Prof., Principal Investigator — University of Cambridge

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03689621/Prot_SAP_000.pdf